CLINICAL TRIAL: NCT05237037
Title: Assessment of Sleep Quality in Patients Utilizing Cannabinoid Therapy
Brief Title: Assessment of Sleep Quality in Cannabinoid Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cerebra Medical (Industry)
Collaborators: Ekosi Health Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: Ekosi
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Poor Sleep Quality
Keywords: Cannabinoid Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The current study aims to assess the impact of starting cannabinoid therapy on sleep quality for individuals with sleep disturbance.

DETAILED DESCRIPTION:
After the initial signing of the consent form, they will complete a battery of baseline questionnaires online on sleep, including the Sleep Regularity Questionnaire, Epworth Sleepiness Scale, Insomnia Severity Index, and the Depression, Anxiety, Stress Scale (DASS-21). That night, before beginning active treatment, participants will be monitored using Cerebra's Level 2 plus ECG system (the Prodigy).

After 6 weeks of active treatment, participants will again complete a night of Level 2 plus ECG recording using the Prodigy, evening, and morning questionnaires, and will repeat baseline sleep questionnaires.

ELIGIBILITY:
Inclusion Criteria

1. A Pittsburgh Sleep Quality Index score >5
2. Between the ages of 40-65
3. No current recreational or medical cannabis use within 4 weeks of the study initiation OR positive urine drug screen (UDS) for Tetrahydrocannabinol
4. No use of anti-psychotics, tricyclic antidepressants, or prescription stimulants
5. No use of medications for promoting sleep (e.g., anti-histamines, benzodiazepines, melatonin).
6. Low risk of Obstructive Sleep Apnea (Low Risk on Berlin Questionnaire), or no presence of moderate or severe Obstructive Sleep Apnea on baseline polysomnography (AHI <15).
7. Has been prescribed THC:CBD combination therapy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have completed standard clinic intake and medical screening at Ekosi Health and been deemed appropriate for a combination THC:CBD treatment will be screened for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Quality (Pittsburgh Sleep Quality Index) | 6 weeks
Change in Objective Sleep Quality (Odds Ratio Product) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ekosi Health Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dzierzewski JM, Donovan EK, Sabet SM. The Sleep Regularity Questionnaire: development and initial validation. Sleep Med. 2021 Sep;85:45-53. doi: 10.1016/j.sleep.2021.06.028. Epub 2021 Jun 28. PMID 34274811
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Lovibond, S.H., & Lovibond, P.F. Manual for the Depression Anxiety Stress Scales. (2nd Ed.) Sydney: Psychology Foundation. (1995).